CLINICAL TRIAL: NCT04871165
Title: Analysis of Immunogenicity, Safety and Efficacy of COVID-19 Vaccines in Immunosuppressed Individuals
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Vilnius University (Other)
Responsible Party: Sponsor
Other Study IDs: OH-VACC-IMMUN
Record Dates: First submitted 2021-04-20; First posted 2021-05-04 (Actual); Last update posted 2022-01-14 (Actual); Status verified 2021-12

CONDITIONS: Hematologic Neoplasms; COVID-19 Vaccines
Keywords: Hematologic Neoplasms; COVID-19 Vaccines; Immunogenicity
MeSH Terms: conditions — Hematologic Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Peripheral blood mononuclear cells, flash frozen lysed white blood cells
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Oncohematological patient group: Patients with prior diagnosis of oncohematological disease vaccinated with SARS-CoV-2 vaccine.
  Interventions: Diagnostic Test: S-binding IgG, RBD-binding IgG and N-binding IgG immunoassays and SARS-CoV-2 serum neutralization assay, quantitative serum immunoglobulin tests; Diagnostic Test: Assessment of proinflammatory cytokine production and immunophenotypic analysis after stimulation with overlapping S-peptides in peripheral blood mononuclear cells (PBMC); Diagnostic Test: Quantitative sequencing for TCR repertoires for SARS-CoV-2-specific antigens
- Healthy control group: Subjects without prior diagnosis of oncohematological disease vaccinated with SARS-CoV-2 vaccine.
  Interventions: Diagnostic Test: S-binding IgG, RBD-binding IgG and N-binding IgG immunoassays and SARS-CoV-2 serum neutralization assay, quantitative serum immunoglobulin tests; Diagnostic Test: Assessment of proinflammatory cytokine production and immunophenotypic analysis after stimulation with overlapping S-peptides in peripheral blood mononuclear cells (PBMC); Diagnostic Test: Quantitative sequencing for TCR repertoires for SARS-CoV-2-specific antigens

INTERVENTIONS:
Diagnostic Test: S-binding IgG, RBD-binding IgG and N-binding IgG immunoassays and SARS-CoV-2 serum neutralization assay, quantitative serum immunoglobulin tests — S-binding IgG, RBD-binding IgG and N-binding IgG immunoassays and SARS-CoV-2 serum neutralization assay, quantitative serum immunoglobulin tests.
Diagnostic Test: Assessment of proinflammatory cytokine production and immunophenotypic analysis after stimulation with overlapping S-peptides in peripheral blood mononuclear cells (PBMC) — Quantitative evaluation of proinflammatory cytokine (IFN-gamma, IL-2 and IL-4) production after stimulation with overlapping S-peptides in peripheral blood mononuclear cells and immunophenotypic analysis (CD45, CD3, CD4, CD8, CD16, CD56, CD14, CD19)
Diagnostic Test: Quantitative sequencing for TCR repertoires for SARS-CoV-2-specific antigens — Quantitative sequencing for TCR repertoires for SARS-CoV-2-specific antigens

SUMMARY:
The study will evaluate the immunogenicity, safety and efficacy of vaccines against severe acute respiratory syndrome corona virus 2 (SARS-CoV-2) in oncohematological patient population and compare the results with patients without prior oncohematological disease. The study is comprised of retrospective and prospective parts. In retrospective part, biobanked residual biological patient material and data will be used. In prospective part, vaccinated oncohematological patients and vaccinated patients without prior oncohematological disease will be invited to participate in long-term follow-up. The subjects will be invited for blood sample collection every three months from the second vaccine dose administration, i.e. 3 mos., 6 mos., 9 mos. etc. When the study subject receives booster dose, additional blood samples for immunogenicity analyses will be collected up to 14 days before and 4-8 weeks after the booster vaccine dose. The follow-up time points occurring every three months will be counted from the last vaccine's dose. Ten time points in total will be collected and tested for humoral and cellular immunogenicity. For safety analysis patient self-documented systemic events (fever, fatigue, headache, chills, vomiting, diarrhea, new or worsened muscle pain, and new or worsened joint pain) occurring up to 7 days following each vaccine dose will be systematized and compared between oncohematological patients and healthy individuals. For efficacy analysis, polymerase chain reaction assay (PCR) confirmed symptomatic disease rates, hospitalization rates and mortality rates will be assessed.

DETAILED DESCRIPTION:
The study will evaluate the immunogenicity, safety and efficacy of vaccines against SARS-CoV-2 in oncohematological patient population and compare the results with patients without prior oncohematological disease. The study is comprised of retrospective and prospective parts. In retrospective part, biobanked residual biological patient material and data will be used. In prospective part, vaccinated oncohematological patients and vaccinated patients without prior oncohematological disease will be invited to participate in long-term follow-up. The subjects will be invited for blood sample collection every three months from the second vaccine dose administration, i.e. 3 mos., 6 mos., 9 mos. etc. When the study subject receives booster dose, additional blood samples for immunogenicity analyses will be collected up to 14 days before and 4-8 weeks after the booster vaccine dose. The follow-up time points occurring every three months will be counted from the last vaccine's dose. Ten time points in total will be collected and tested for humoral and cellular immunogenicity, detailed below.

The study sample size is based on the number of oncohematological patient population, eligible for vaccination. Our assumed study sample size during the whole study period is up to 2500 adult patients + up to 200 adolescent patients with oncohematological disease and up to 500 adult + up to 70 adolescent patients without prior oncohematological disease. The size of the control group is aimed at achieving sufficient samples for statistical comparison of the groups. All study participants will have received a vaccination schedule specified in each vaccine's Summary of Product Characteristics.

For humoral immunogenicity evaluation blood serums from up to 2500 adult patients + up to 200 adolescent patients with oncohematological disease and up to 500 adult + up to 70 adolescent patients without prior oncohematological disease will be tested at the following time points: 1) up to 10 days before the first vaccine dose, 2) on the day of second vaccine dose, 3) 1 to 3 weeks after second vaccine dose. Further samples will be obtained every 3 months after administration of second vaccine dose. When the study subject receives booster dose, additional blood samples for immunogenicity analyses will be collected up to 14 days before and 4-8 weeks after the booster vaccine dose. The follow-up time points occurring every three months will be counted from the last vaccine's dose. 10 follow-up time points in total. The samples will be used to perform S-binding immunoglobulin G (IgG), receptor-binding domain (RBD)-binding IgG and N-binding IgG immunoassays, SARS-CoV-2 serum neutralization assay against different SARS-CoV-2 variants and quantitative serum immunoglobulin tests.

For cellular immunogenicity evaluation PBMC samples from up to 100 oncohematological patients and 20 healthy individuals will be tested at the following time points: 1) up to 10 days before the first vaccine dose and 2) 1 to 3 weeks after second vaccine dose. Further samples will be obtained every 3 months after administration of second vaccine dose. When the study subject receives booster dose, additional blood samples for immunogenicity analyses will be collected up to 14 days before and 4-8 weeks after the booster vaccine dose. The follow-up time points occurring every three months will be counted from the last vaccine's dose. Ten follow-up time points in total. Cellular immunogenicity will be evaluated in oncohematological patients, who may have a weak humoral response to vaccines. The following groups of oncohematological patients will be included: 1) 20 to 40 recent recipients of allogeneic stem cell transplantation (allo-SCT), meeting these requirements: 2-8 months after allo-SCT; cluster of differentiation 3 (CD3) positive cell count >0.1*109/L; patients with mild chronic graft-versus-host disease (GvHD) and/or receiving <0.5mg/kg prednisolone (or equivalent); patients with <2nd grade acute GvHD; >3 months after anti-CD20 therapy; postgraft immunosuppression with calcineurin inhibitors is allowed; 2) 20 to 40 patients after recent administration of proteasome inhibitors (0-30 days after treatment), who received at least one full cycle of treatment and achieved a satisfactory and stable disease response, allowing a safe temporary treatment discontinuation for immunization against COVID-19; 3) 20 to 40 patients after a recent anti-CD20 administration (0-180 days after treatment), who received at least one full cycle of treatment and achieved satisfactory and stable disease response, allowing a safe temporary treatment discontinuation for immunization against COVID-19. Other specific patient groups will be enrolled in the cellular immunogenicity part, as the primary analysis results show which specific subpopulations lack humoral immune response. PBMC samples from individuals without prior diagnosis of oncohematological disease will be selected randomly. The samples will be used for assessment of proinflammatory cytokine (interferon-gamma (IFN-gamma), interleukin-2 (IL-2) and IL-4) production and immunophenotypic analysis (CD45, CD3, CD4, CD8, CD16, CD56, CD14, CD19) after stimulation with overlapping S-peptides in PBMC.

Cellular immunogenicity will be evaluated by performing quantitative sequencing for T-cell receptor (TCR) repertoires for SARS-CoV-2-specific antigens using immunoSEQ technology (Adaptive Biotechnologies Inc., 1165 Eastlake Ave E, Seattle, Washington 98109, United States).

For safety analysis patient self-documented systemic events (fever, fatigue, headache, chills, vomiting, diarrhea, new or worsened muscle pain, and new or worsened joint pain) occurring up to 7 days following each vaccine dose will be systematized and compared between oncohematological patients and healthy individuals.

For efficacy analysis, PCR confirmed symptomatic disease rates, hospitalization rates and mortality rates will be assessed. In case of detected breakthrough infection, additional biological samples will be obtained as soon as possible to evaluate humoral and cellular immunity at the time of infection and repeated until PCR-negativity is achieved.

ELIGIBILITY:
Inclusion criteria for oncohematological patients

1. >/= 12 years of age.
2. Prior diagnosis of oncohematological disease.
3. The patient has signed an informed consent form.
4. The patient was vaccinated with SARS-CoV-2 vaccine.

Inclusion criteria for healthy individuals

1. >/= 12 years of age.
2. Patients without prior diagnosis of oncohematological disease.
3. The patient has signed an informed consent form.
4. The patient was vaccinated with SARS-CoV-2 vaccine.

Exclusion criteria No exclusion criteria will be applied.

Min Age: 12 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: Patients with haematological malignancies compared to healthy control group.
Sampling Method: Non-Probability Sample
Enrollment: 3270 (Estimated)
Dates: Start 2021-03-24 (Actual); Primary Completion 2024-03-01 (Estimated); Study Completion 2024-03-01 (Estimated)

PRIMARY OUTCOMES:
Humoral immune response elicited by COVID-19 vaccines | 7 to 21 days after the second vaccine dose
  SARS-CoV-2 antibody level in response to COVID-19 vaccines

SECONDARY OUTCOMES:
Cellular immune response elicited by COVID-19 vaccines | 7 to 21 days after the second vaccine dose
  Evaluation of T-cell phenotype and cytokine production after stimulation with overlapping S-peptides in peripheral blood mononuclear cells using flow cytometry in response to COVID-19 vaccines; Quantitative sequencing for TCR repertoires for SARS-CoV-2-specific antigens
Safety of COVID-19 vaccines | up to 7 days after each vaccine dose administration
  Number of systemic events (fever, fatigue, headache, chills, vomiting, diarrhea, new or worsened muscle pain, and new or worsened joint pain)
Efficacy of COVID-19 vaccines | starting 7 days after the completion of vaccination schedule and up to 100 weeks
  Evaluation of COVID-19 incidence

CONTACTS AND LOCATIONS:
Locations (1):
- Vilnius University Hospital Santaros Klinikos, Vilnius, Lithuania

IPD SHARING:
Plan to Share IPD: No
No individual data will be shared

REFERENCES:
- [Derived] Maneikis K, Sablauskas K, Ringeleviciute U, Vaitekenaite V, Cekauskiene R, Kryzauskaite L, Naumovas D, Banys V, Peceliunas V, Beinortas T, Griskevicius L. Immunogenicity of the BNT162b2 COVID-19 mRNA vaccine and early clinical outcomes in patients with haematological malignancies in Lithuania: a national prospective cohort study. Lancet Haematol. 2021 Aug;8(8):e583-e592. doi: 10.1016/S2352-3026(21)00169-1. Epub 2021 Jul 2. PMID 34224668